CLINICAL TRIAL: NCT04827043
Title: Ultrasound Guided Quadratus Lumborum Block Versus Thoracic Paravertebral Block in Gynacological Cancer Surgery
Brief Title: Quadratus Lumborum Block Versus Thoracic Paravertebral Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fatma Gomaa Hussein, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Quadratuslumborum block & TPVB
Record Dates: First submitted 2021-03-09; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Analgesia
Keywords: Quadratus lumborum block; Thoracic paravertebral block; Postoperative analgesia

STUDY DESIGN:
Intervention Model Description: A prospective randomized comparative study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After approval of The InstitutionalEthics Committee of The National Cancer Institute ,Cairo University, 50 patients scheduled for gynacological cancer surgery will be enrolled in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block (Experimental): QLB group: will receive 0.3ml/Kg bupivacaine 0.25% ( keeping in mind not to exceed the maximum recommended toxic dose of plain bupivacaine which is 2.5 mg/Kg & 3mg/Kg with epinephrine), single injection sonar guided.
  Interventions: Combination Product: Ultrasound guided quadratus lumborum block
- Thoracic paravertebral block (Experimental): PVB group: will receive 0.25ml/Kg/side of 0.375% bupivacaine with epinephrine 5ug/ml, yielding the same dose of bupivacaine of 1.875mg/ml at the level of T10 as a single injection sonar guided.
  Interventions: Combination Product: Ultrasound guided thoracic paravertebral block

INTERVENTIONS:
Combination Product: Ultrasound guided quadratus lumborum block — prospective randomized comparative study between Group (1) : quadratus lumborum block
  Other Names: QLB
  Arms: Quadratus lumborum block
Combination Product: Ultrasound guided thoracic paravertebral block — PVB group: will receive 0.25ml/Kg/side of 0.375% bupivacaine with epinephrine 5ug/ml, yielding the same dose of bupivacaine of 1.875mg/ml at the level of T10 as a single injection sonar guided.
  Other Names: PVB
  Arms: Thoracic paravertebral block

SUMMARY:
This study is to assess and compare the analgesic efficacy and safety of quadratus lumbotum block and paravertebral block in gynacological cancer patients.

DETAILED DESCRIPTION:
All patients will be medically checked in the preoperative assessment clinic {history, physical examination, investigations (e.g. complete blood picture, coagulation profile , liver & kidney functions , ECG for patient above 40 years, chest x-ray for patients above 60 years and any other necessary investigations required for risky patients. ) }.

The patients will be randomly allocated into two equal groups(25 patients for each group) with a computer-generated list (www.Random.org).

QLB group: will receive 0.3ml/Kg bupivacaine 0.25% ( keeping in mind not to exceed the maximum recommended toxic dose of plain bupivacaine which is 2.5 mg/Kg & 3mg/Kg with epinephrine).

PVB group: will receive 0.25ml/Kg/side of 0.375% bupivacaine with epinephrine 5ug/ml, yielding the same dose of bupivacaine of 1.875mg/ml at the level of T10.

* In the recovery room, the patients will be continuous monitored for pulse, blood pressure, oxygen saturation.
* Humidified oxygen 3L/min. by nasal prong will be delivered to all patients.
* Portable ultrasound machine , nerve stimulator, pressure injector monitor ,resuscitation equipment &drugs (e.g. epinephrine, lipid emulsion ), sterile gloves and surgical towels should be available.
* Intravenous(IV) 18 gauge cannula will be inserted. Midazolam 0.02 mg/Kg will be administered.

While the patients in the supine or lateral position, they will receive bilateral single injection ultrasound guided QLBs under complete sterilization of the abdomen with sterile solution (iodine povacryl & isopropyl alcohol solution). All patients will be monitored throughout the performance of the block & all data will be recorded. A linear ultrasound transducer probe (6-13MHZ), or curved probe (according to patients BMI). ( Sonosite M-turbo; Inc., Bothell, WA, USA) in a sterile cover will be placed at the level of the anterosuperior iliac spine and moved cranially until the three muscle layers of the abdomen will be identified: external oblique, internal oblique, and transversus abdominis muscles. The external oblique muscle will be followed posterolaterally until its posterior border visualize (hook sign) leaving underneath the internal oblique muscle, like a roof over the QL muscle. The probe will be tilted down to identify a bright hyperechoic line that corresponded with the intermediate layer of the thoracolumber fascia(Blanco et al.,2015).

A 21 gauge blunt, insulated, echogenic needle will be inserted in plane . The optimal point of injection will be determined using hydrodissection (3-5 mL normal saline). The site of the needle will be confirmed in place by ultrasound guided, nerve stimulator (B- Braun) & pressure injector monitor.

After negative aspiration, we will inject 0.3mL/Kg bupivacaine 0.25% in each side in QLB group. The patients will be monitored for about 20-30 minutes before induction of anesthesia.

While the TPVB will be performed by single injections at the level of T10 vertebra. The patients will be placed in the sitting position, and the spinal process of T10 will be palpated. Then a linear ultrasound transducer probe (6-13 MHZ).

( Sonosite M-turbo; Inc., Bothell, WA, USA) in a sterile cover will be placed at the corresponding transverse process to be clearly visualized and the skin-transverse process distance will be measured on both sides. After infiltration of the skin and subcutaneous tissue with 1% lidocaine with epinephrine 5ug/ml, an 18G Touphy needle will be inserted perpendicular to the skin, approximately 2.5 cm from midline, until contact with the transverse process will be established ( It is important to visualize the pleura very clearly at all times ). The needle will then slightly withdrawal & reinserted 1-1.5 cm deeper either caudally or cranially for the transverse process (TP). The site of the needle will be confirmed in place by ultrasound guided, nerve stimulator (B- Braun) & pressure injector monitor.

After careful aspiration, patients will be received a slow injection of 0.25mL/Kg/side of 0.375% bupivacaine with epinephrine 5ug/ml at the level of T10. The patients will be monitored for about 30 minutes before induction of anesthesia. Induction of general anesthesia will be done.

After full awakening from anesthesia, the patient will be transferred to the recovery room. In the recovery room, the patient will be continuous monitored & humidified oxygen will be applied for about 1 hour. Then a standardized analgesic regimen consisting of regular IV/oral paracetamol 1g every 6 hours combined with PCA morphine (on demand) will be initiated. Patients required additional analgesia will be received IV ketorolac(15-30mg).

A trained anesthetist not involved in the study & blinded to the patient group will measure the VAS, morphine requirements & patient satisfaction.

ELIGIBILITY:
1. Inclusion criteria

1. ASA I-III.
2. Age ≥ 20 & ≤ 70
3. Body mass index (BMI): Less than forty and more than twenty.
4. Patients undergoing major gynacological cancer surgeries.

2. Exclusion criteria

1. Patient refusal.
2. History of sensitivity to local anesthetic (amide group).
3. History of psychological disorders.
4. Coagulopathies: hereditary (e.g. hemophilia, fibrinogen abnormalities& deficiency of factor II) - acquired (e.g. liver disease, vitamin K deficiency & therapeutic anticoagulants drugs).
5. Localized infection.
6. Morbid obese BMI>40.
7. Incooperative patients.
8. Patients on chronic pain therapy.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Baseline pain till first 24 hours postoperative
  Pain score will be measured according to severity

SECONDARY OUTCOMES:
Morphine demands postoperative | First 24 hours postoperative
  The amount of morphine required to relieve pain will be recorded
Patient satisfaction | First 24 hours postoperative
  Patient satisfaction measured by visual analogue score

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A El-samahy, Professor, Study Director — National Cancer Institute (NCI); Ekramy M Abd-elghaffar, MD, Study Director — National Cancer Institute (NCI); Esam Ab Mahran, MD, Study Director — National Cancer Institute (NCI)

IPD SHARING:
Plan to Share IPD: Yes
Starting in April 2021 Ending in July 2021
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately after publication No end date
Access Criteria: Any one who wishes to access the data
URL: http://www.scopus.com

REFERENCES:
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488